CLINICAL TRIAL: NCT02309996
Title: A Supervisor Training Program for Work Disability Prevention: A Cluster RCT
Brief Title: SMART Supervisor Training Program to Prevent Work Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lakehead University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Liberty Mutual Research Institute for Safety (Industry); Institute for Work & Health (Unknown)
Responsible Party: Principal Investigator, Vicki Kristman, Assistant Professor, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOP-130505
Record Dates: First submitted 2014-12-02; First posted 2014-12-05 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Work Disability Reduction and Prevention; Improving Return-to-Work Outcomes
Keywords: Randomized Controlled Trial; Intervention Studies; Inservice Training; Personnel Management; Work place; Work accommodation; Job modification; Supervision; Administration; Return to Work; Industrial Psychology; Human Engineering; Risk Management; Organization and Administration; Work Disability; Occupational Diseases; Occupational Injury; Occupational Health; Occupational Exposure; Sick Leave; Absenteeism; Employee Health
MeSH Terms: conditions — Occupational Diseases; Occupational Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervisor Training Program (Experimental): All supervisors from work units randomized to the intervention will receive a supervisor training program, the Supervisor/Manager Accommodation Recognition & Training (SMART) Program. This training program is modeled on a program developed by Shaw and colleagues of the Liberty Mutual Research Institute for Safety (LMRIS). The aim of the training program is to prevent/reduce work disability by improving supervisor communication, response to workplace injury, and problem solving mechanisms. The training program is designed to be administered by two facilitators to groups of 10 to 12 supervisors, during one 4-hour session or two 2-hour sessions. The training program delivery mode includes PowerPoint presentation with supplementary audio or video segments, case studies, and group discussion.
  Interventions: Behavioral: Supervisor Training Program
- No Supervisor Training Program (No Intervention): All supervisors from work units randomized to the control group will not receive the supervisor training program.

INTERVENTIONS:
Behavioral: Supervisor Training Program
  Arms: Supervisor Training Program

SUMMARY:
Supervisors of injured workers play a key role in preventing prolonged work absences. Providing supervisors with tools to improve their response to musculoskeletal and other workplace injuries or illnesses may improve worker health and disability outcomes.

The primary objective of this research study is to determine the effectiveness of the supervisor training program, the SMART Supervisor Training Program, on reducing the total duration of workers' lost-time claims. The secondary objectives are 1) to determine the effectiveness of the training program on reducing the cumulative incidence of workers' lost-time injuries and sick leave days; 2) to determine if implementation of the training program is associated with improvements in hypothesized mediating variables, such as attitudes toward job accommodations, response to workplace injury, and communication with employees and healthcare providers; 3) to investigate the implementation of the training program by conducting a process evaluation.

The investigators hypothesize that:

1. the duration of lost-time claims for workers working under supervisors receiving the training program will be shorter than the duration of lost-time claims for workers with supervisors in the control group;
2. the cumulative incidence of lost-time injuries and sick leave days will be lower in the group receiving the training program compared to the control group;
3. the training program will be associated with increased knowledge, response, communication and changed attitudes towards workplace accommodation.

This research is of significance to North American employers and compensation systems because there is a lack of knowledge about the usefulness of supervisor training to prevent or reduce work disability. It also has important implications for guiding employer policies and practices, and for identifying circumstances where supervisor training should be a priority.

DETAILED DESCRIPTION:
This study is a multi-centred, cluster randomized, controlled, single-blinded, fixed sample trial.

The project will involve several large Canadian and American employers. Participating work units within the organizations will be randomly assigned to either the training program (intervention group) or not (control group). Randomizing geographically separate work units works best to prevent contamination of supervisors selected to be the control group. However, the employer will decide what constitutes a work unit (e.g., separate building, division, etc.). The work units will be pair-matched into clusters based on number of employees, gender proportions, and work tasks as best as possible. A total of 86 work units (43 work unit pairs) including approximately 350 supervisors is required to achieve the primary objective, with fewer work units and supervisors required to achieve the secondary objectives. Within each cluster, one work unit will receive the training program and the other will act as the control. All supervisors within those work units randomized to receive the intervention will attend a four-hour supervisor training session. Before training is administered to the randomly assigned work units, all supervisors (intervention group and control group) will receive an email with an attached information pamphlet about principles for successful return to work. The purpose of the information pamphlet is to minimize the Hawthorne Effect, whereby subjects change their behaviour in response to the knowledge that they are being studied or monitored.

The work disability outcomes (duration of lost-time injuries in days, and cumulative incidence of lost-time injuries and sick leave days) will be determined from workplace records, and outcomes data will be extracted and analyzed at the level of the work unit. Since the intervention is a training program, it is impossible to blind the participating supervisors. However, the data extractor and individuals working in each employer's Occupational Health & Safety Department will be blinded to the results of the work unit randomization and no other workers will be informed if the supervisors in their work unit received the training program or not.

To collect information about the hypothesized mediating variables, consenting supervisors will be asked to complete three online questionnaires: baseline and two follow-up questionnaires (three and six months post-randomization). The baseline and follow-up questionnaires will also collect information on potential moderating and confounding factors including workplace safety culture, supervisor autonomy, corporate disability management, leadership style, workplace social capital, and workers' physical work demands, supervisor demographics, and characteristics of supervised workers (e.g., number, gender proportions, unionization status). Analysis of the mediating variables will be conducted at the level of the work unit. Data for the process evaluation will be obtained from a brief exit training program evaluation survey distributed to participants in the intervention group as well as the three and six month follow-up questionnaires.

This is a pragmatic, intent-to-treat trail, so participants will be analyzed according to the group they were randomly assigned to. However, the investigators will also obtain information about supervisor transfers among work units (and the direction of the transfers) for the one year period post-randomization to understand how such transfers may have influenced the results.

ELIGIBILITY:
Inclusion Criteria:

* Supervisors
* Currently employed at the work units selected by participating employers
* Supervise at least one working employee (i.e., non-supervisor)
* Would deal with issues of work accommodation should the need arise

Exclusion Criteria:

* Higher level supervisors who only supervise lower-level supervisors
* Do not speak/read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2014-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Total duration of workers' lost-time claims due to injury or illness for existing and new claims | 1 year period post-randomization
  Aggregated lost-time due to injury or illness.

SECONDARY OUTCOMES:
Cumulative incidence of workers' lost-time injuries | 1 year period post-randomization
  Summing all new cases of lost-time injuries across worker groups..
Total number of workers' sick leave days | 1 year period post-randomization
  Summing up sick leave days across worker groups.
Job Accommodation Scale (JAS) | Baseline, 3 months, 6 months
  The JAS is a 21-item self-report measure developed to assess the likelihood that various job modification might be supported in the workplace. For more information see:
  W. S. Shaw, V. L. Kristman, K. Williams Whitt, S. Soklaridis, Y. Huang, P. Côté and P. Loisel. 2014. The Job Accommodation Scale (JAS): psychometric evaluation of a new measure of employer support for temporary job modifications. Journal of Occupational Rehabilitation 24 (4): 755-765.
Supervisor's Role in Rehabilitation Questionnaire | Baseline, 3 months, 6 months
  This instrument asks supervisors to rank their self-efficacy to engage in all of the rehabilitation tasks associated with vocational rehabilitation. The survey uses a series of Likert scales, using response categories which classify each rehabilitation task as either being: "very difficult to do"; "hard to do"; "easy to do"; or "very simple to do". This scale is seen as a continuum of supervisor ability, and a measure of their self-rated capacity to engage in vocational rehabilitation at their own workplaces. The reliability estimate for the use of this rating scale is acceptable (Cronbach alpha = 0.89) and Rasch analysis supports the premise that all 20 rehabilitation items being estimated are unidimensional.
  I. Blackman and K. Chiveralls. 2011. Factors influencing workplace supervisor readiness to engage in workplace-based vocational rehabilitation. Journal of Occupational Rehabilitation 21 (4): 537-546.
Behaviour Measure for Supervisors to Support Return to Work (SSRW) questionnaire | 6 months
  The SSRW was developed using supervisor and employee populations and there is a version for supervisors and a version for employers. The 42 items in the scale are related to supervisor behaviours during an employee's absence from work and subsequent return to work. The measure consists of four sub-scales: communication and support during sick leave, inclusive behaviour upon initial return, negative behaviours and general proactive support following return to work. A total score is obtained by summing the responses, with a higher score indicating more supportive behaviours. The measure has good internal consistency, test-retest reliability, and construct validity. The SSRW will be included in the 6-month follow-up questionnaire only.
  F. Munir, J. Yarker, B. Hicks and E. Donaldson Feilder. 2012. Returning employees back to work: developing a measure for Supervisors to Support Return to Work (SSRW). Journal of Occupational Rehabilitation 22 (2): 196-208.
Supervisor Support Scale from the "Readiness for RTW Study" | Baseline, 3 months, 6 months
  The supervisor support scale was designed to assess the relations between injured workers and supervisors. This scale is based on items from a previously used questionnaire and also includes items developed by a clinical psychologist, organizational psychologist, psychometrist, and a graduate student in community health. Although this scale was originally developed for response by injured workers, we modified the 8-item scale for supervisor response. We will average all responses not indicating "Don't Know" to determine a supervisor support score from 1 to 4 where higher scores indicate better supervisor interaction.
  R. Franche, C. N. Severin, S. Hogg Johnson, H. Lee, P. Côté and N. Krause. 2009. A multivariate analysis of factors associated with early offer and acceptance of a work accommodation following an occupational musculoskeletal injury. Journal of occupational and environmental medicine 51 (8): 969-983.
Supervisory Behavior Questionnaire | Baseline, 3 months, 6 months
  The supervisory behaviour scale was designed to assess positive supervisory behaviour regarding communication with the employee, promotion of gradual return to work, and consultation with other professionals. The scale includes 7 statements about interactions between supervisors and injured workers and asks supervisors to indicate how much they agree or disagree with each statement. Responses to all statements will be summed and will result in a final score between 7 and 35 where lower scores indicate positive supervisor behaviour.
  K. Nieuwenhuijsen, J. H. Verbeek, A. G. de Boer, R. W. Blonk and F. J. van Dijk. 2004. Supervisory behaviour as a predictor of return to work in employees absent from work due to mental health problems. Occupational and Environmental Medicine 61 (10): 817-823.
Supervisor and Healthcare Provider Interactions questionnaire | Baseline, 3 months, 6 months
  Communication with healthcare providers will be measured with a questionnaire assessing supervisors' interactions with healthcare providers developed specifically for the mixed-methods study. The five questions were selected from existing publications as we could not find an existing scale appropriate for our needs through the literature review. Three constructs will be measured from these questions including healthcare communication (i.e., do you communicate with providers?), healthcare beliefs (i.e., does the supervisor believe the provider understands the nature of the job?), and healthcare information (i.e., how often does a provider help you return a worker to work?). The scale has good face validity and reliability in the supervisor population as determined from our previous project.
Global Work Safety Climate (GWSC) Scale | Baseline, 6 months
  A 6-item measure that assesses global work safety climate. For more information:
  S.E. Hahn. 2008. A short scale for measuring safety climate. Safety science 46 (7): 1047-1066.
Organizational Policies and Practices (OPP) Scale (13 questions about organizational disability management policies and practices) | Baseline
  Amick BC III, Habeck RV, Hunt A, et al. Measuring the impact of organizational behaviors on work disability prevention and management. Journal of Occupational Rehabilitation 10 (1): 21-38.
Supervisor Autonomy for Provision of Job Accommodations questions | Baseline
  Three questions using a likert scale.
Leader Behavior Description Questionnaire (LBDQ) | Baseline, 3 months
  Halpin AW. Manual for the Leader Behaviour Description Questionnaire. Columbus, OH:Bureau of Business Research, Ohio State University, 1957.
Physical Workload Questionnaire (PWQ) | Baseline
  Bot SDM, Terwee CB, van der Windt DAWM, et al. Internal consistency and validity of anew physical workload questionnaire. Occupational and Environmental Medicine 2004;61:980-86.
Training program reach (proportion of the target group that participates) | Up to 1 month post-randomization
  Calculation of the percentage of supervisors that participate in the training.
Training program dose delivered (efforts of the trainers) | Up to 1 month post-randomization
  Training program dose delivered (efforts of the trainers).
Training program dose received (extent to which the supervisors have followed the training) | Up to 1 month post-randomization
  Training program dose received (extent to which the supervisors have followed the training).
Training program fidelity (extent to which the training program was delivered according to the protocol) | Up to 1 month post-randomization
  Training program fidelity (extent to which the training program was delivered according to the protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki L Kristman, PhD, Principal Investigator — Lakehead University
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada